CLINICAL TRIAL: NCT04442893
Title: Exploring the Effect of Rumination-Focused Cognitive Behaviour Therapy on Depressive Symptoms in Patients With Schizophrenia: A Randomized Controlled Trial
Brief Title: Exploring the Effect of Rumination-Focused Cognitive Behaviour Therapy in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Bali Psychiatric Center (Other)
Responsible Party: Principal Investigator, Chiu-Yueh Yang, Associate Professor, Nursing Department, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YM108038F
Record Dates: First submitted 2019-09-02; First posted 2020-06-23 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Randomized Controlled Trial
Keywords: Rumination-Focused Cognitive Behaviour Therapy(RFCBT); depressive symptom; Schizophrenia
MeSH Terms: conditions — Depression; Schizophrenia

STUDY DESIGN:
Intervention Model Description: The participants were divided into experimental and control groups through block randomization
Who Masked: Participant
Masking Description: The data of PANSS were collected by a research assistant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group would be provided with a 6- session RFCBT program for 12 weeks (60-90 mins, once every two weeks).
  Interventions: Behavioral: Rumination-Focused Cognitive Behaviour Therapy
- Control group (Other): The control group would receive a 6- session Health Education program for 12 weeks (60-90 mins, once every two weeks)
  Interventions: Other: Health Education programme

INTERVENTIONS:
Behavioral: Rumination-Focused Cognitive Behaviour Therapy — Rumination-Focused Cognitive Behavioural Therapy(RFCBT) is based on a differentiation between functional and dysfunctional styles of perseverative thinking with the helpful style characterized as a concrete, process-focused and specific style of thinking and the idea that rumination is a habit maintained by negative reinforcement. In line with the theoretical assumptions, RFCBT combines strategies from behavioral activation with strategies to foster concrete, process-focused and specific thinking.
  Arms: Experimental group
Other: Health Education programme — Health education programme would be any planned activity or set of activities aimed at increasing health literacy and developing life skills conducing to health (e.g. decision making, problem solving, critical thinking, interpersonal skills, stress management, coping with emotions).
  Arms: Control group

SUMMARY:
This study will explore the effect of Rumination-Focused Cognitive Behaviour Therapy on depressive symptoms in patients with schizophrenia for three months. A randomized controlled trial is conducted in a psychiatric center in northern Taiwan. All participants are randomized to two groups using blocked randomization. The experimental groups are provided with a 6- session RFCBT program for 12 weeks (60-90 mins, once every two weeks), while the control groups receive a 6- session Health Education program for 12 weeks (60-90 mins, once every two weeks). All participants who suffered from depressive symptoms at both baseline and 3-month follow-up will be evaluated using the Beck Depression Inventory(BDI-II), Chinese Response Style Questionnaire-short form revised(CRSQ-10), Internalized Stigma of Mental Illness (ISMI) Scale, and Herth Hope Index Chinese Version(HHI).

DETAILED DESCRIPTION:
Background:

Depressive symptoms are one of the core symptoms in patients with schizophrenia, but the effect of depressive symptoms on patients is easily overlooked. Severe depressive symptoms in patients with schizophrenia are not only affecting the quality of life but also the risk factors of suicide.

Aim:

The investigators hypothesize that Rumination-Focused Cognitive Behaviour Therapy(RFCBT) could have significant effect of depressive symptoms. Therefore, in this study, the investigators will explore the effect of Rumination-Focused Cognitive Behaviour Therapy(RFCBT) on depressive symptoms in patients with schizophrenia.

Methods:

The study is conducted as a two-arm, single-blinded, randomized controlled trial in a psychiatric center in northern Taiwan. Participants are randomly allocated in a 1:1 ratio to two groups using blocked randomization. The experimental groups are provided with a 6- session RFCBT program for 12 weeks (60-90 mins, once every two weeks), while the control groups receive a 6- session Health Education program for 12 weeks (60-90 mins, once every two weeks) .

Participants and demographic data:

Participants who have been diagnosed with schizophrenia according to DSM-IV criteria took part in the study after informed consent is obtained. All participants are 20 years of age or older and are receiving a stable dosage of antipsychotics, and have no history of cognitive impairment. The participants are able to express themselves and to individually complete the Beck Depression Inventory(BDI-II), Chinese Response Style Questionnaire-short form revised(CRSQ-10), Internalized Stigma of Mental Illness (ISMI) Scale, and Herth Hope Index Chinese Version(HHI).

Measures:

The demographic characteristics include five continuous variables (age, age at onset, duration of disease, years of education, chlorpromazine equivalent dose (Andreasen, Pressler, Nopoulos, Miller, & Ho, 2010) and four categorical variables (sex, marital status, work status, antidepressants).

Procedure and Data collection:

All procedures are approved by both national Ying Ming university(IRB YM108038F) and the psychiatric center (IRB 1080009-01). Following informed consent, each participant will fill out a demographic questionnaire and complete the BDI-II, CRHQ-10, ISMIS, and HHI once at baseline and twice an interval of three months. A well-trained and licensed psychiatric nurse will perform the data collection and assists the participants if there were difficulties reading or understanding the questionnaires.

Statistical analysis:

This study will employ Predictive Analytics Suite Workstation (IBM SPSS 24.0) to analyze the collected data. The data analyses will include demographic variables and the scores of BDI-II, CRHQ-10, ISMIS, and HHI at the interval of three months of all of the participants.

ELIGIBILITY:
Inclusion Criteria:

* The participants are diagnosed with schizophrenia by Diagnostic and Statistical Manual of Mental Disorders, Five Edition (DSM-V), an age of between 20 and 65 years, hospitalization in a rehabilitation unit, and a stable condition at the time of data collection.
* The participants are able to provide written informed consent and comprehend the instruments.
* The participants consent to receive a 6- session RFCBT program or a 6- session Health Education program and complete a package of questionnaires.
* The participants are satisfied the screening criteria including the Positive and Negative Syndrome Scale (PANSS) for positive syndromes < 5, the Mini-Mental State Examination (MMSE) ≥ 24, and the Brief Symptom Rating Scale (BSRS-5) ≥ 6.

Exclusion Criteria:

* The participants who have intellectual disturbances (organic mental disorders) or substance abuse issues through a chart review.
* The participants who are not willing to sign the consent.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Yueh Yang, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 44 | 41
Completed | 34 | 36
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.18 (7.88) | 51.24 (8.09) | 51.21 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 23 | 19 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of disease [Mean (Standard Deviation); unit: years] | 29.05 (8.43) | 26.73 (8.68) | 27.93 (8.58)
CPZ equivalent doses [Mean (Standard Deviation); unit: mg] — It represents the amount of a given drug equivalent to CPZ 100 mg.
  mg | 503.77 (260.58) | 471.29 (286.56) | 488.11 (272.26)
Year of Education [Mean (Standard Deviation); unit: years] | 11.68 (2.88) | 11.39 (2.91) | 11.54 (2.89)
Marital status [Count of Participants; unit: Participants]
  Single | 36 | 35 | 71
  Married | 8 | 6 | 14
Religious preference [Count of Participants; unit: Participants]
  None | 5 | 8 | 13
  Buddha/Christian/other | 39 | 33 | 72
Work status [Count of Participants; unit: Participants]
  Not employed | 33 | 26 | 59
  Employed | 11 | 15 | 26
Antidepressant users [Count of Participants; unit: Participants] — This is defined as the number of participants who using antidepressant.
  Participants
    No | 39 | 34 | 73
    Yes | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory (BDI-II)
Description: The Beck Depression Inventory-II (BDI-II) is a 21-item self-report depression screening measure. Each item is rated on a four-point Likert-type scale ranging from 0 to 3, which with possible scores ranging from 0 to 63. The BDI-II has been translated into a Chinese version. Higher total scores indicate more severe depressive symptoms, and a score of >16 points is considered suggestive of the presence of clinically significant depressive symptom intensity.
  In this study, the investigators will explore the change of BDI-II score among baseline, after intervention and three-month follow-up.
Time Frame: For two study groups, the measure time points are at baseline(T0), after intervention (T1) and three-month follow-up (T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 44 | 41
score on a scale
  T0 | 16.89 (12.32) | 16.88 (14.63)
  T1 | 16.60 (10.80) | 18.70 (12.88)
  T2 | 15.56 (11.26) | 23.03 (14.81)

2. Primary Outcome: Chinese Response Style Questionnaire-short Form Revised (CRSQ-10)
Description: The Chinese Response Style Questionnaire-short form revised (CRSQ-10) is a self-report measure of rumination, comprising ten items and describing the factors of brooding and reflection. Each item is rated on a four-point Likert-type scale ranging from 1 (strongly disagree) to 4 (strongly agree), which with possible scores ranging from 10 to 40. The CRSQ-10 has been used to evaluate the intensity of ruminative responses to depressed mood.
  In this study, the investigators will explore the change of CRSQ-10 score among baseline, after intervention and three-month follow-up.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 44 | 41
score on a scale
  T0 | 26.25 (6.75) | 26.51 (6.62)
  T1 | 26.46 (5.77) | 26.68 (5.44)
  T2 | 27.38 (5.64) | 25.33 (5.01)

3. Secondary Outcome: The Internalized Stigma of Mental Illness (ISMI) Scale
Description: The Internalized Stigma of Mental Illness (ISMI) Scale is a 29-item self-report questionnaire measuring self-stigma among persons with psychiatric disorders. Each item is rated on a four-point Likert scale from 1 (strongly disagree) to 4 (strongly agree), which with possible scores ranging from 29 to 116. The ISMI Scale has been translated into a Chinese version. Higher scores indicating greater self-stigma.
  In this study, the investigators will explore the change of ISMI Scale score among baseline, after intervention and three-month follow-up.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 44 | 41
score on a scale
  T0 | 71.86 (11.33) | 68.63 (11.53)
  T1 | 71.52 (12.43) | 70.35 (10.29)
  T2 | 69.12 (12.83) | 70.44 (10.08)

4. Secondary Outcome: Herth Hope Index Chinese Version(HHI)
Description: The Herth Hope Index (HHI) comprises 12-item self-report measure of hopefulness. Each item is rated on a four-point Likert scale from 1 (strongly disagree) to 4 (strongly agree), which with possible scores ranging from 12 to 48. The HHI has been translated into a Chinese version. Higher scores indicating greater hopefulness.
  In this study, the investigators will explore the change of HHI score among baseline, after intervention and three-month follow-up.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 44 | 41
score on a scale
  T0 | 33.86 (6.23) | 33.54 (4.35)
  T1 | 35.00 (6.35) | 32.62 (6.09)
  T2 | 34.71 (6.62) | 32.17 (6.81)

ADVERSE EVENTS:
Time Frame: 24weeks
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 0/44 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT04442893/Prot_SAP_000.pdf